CLINICAL TRIAL: NCT05989867
Title: Evaluation of Oral Glucose Tolerance Testing in Patients With Post-pancreatitis Diabetes Mellitus for Diagnosis and Characterization: a Cross-sectional Trial
Brief Title: Evaluation of OGTT in Patients With Post-pancreatitis Diabetes Mellitus for Diagnosis and Characterization
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, professor, Changhai Hospital
Other Study IDs: ESTABLISH
Record Dates: First submitted 2023-07-10; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Chronic Pancreatitis; Pancreatogenic Type 3C Diabetes Mellitus; Diabetes Mellitus; Oral Glucose Tolerance Test
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CP: patients with chronic pancreatitis but not combined with diabetes
  Interventions: Diagnostic Test: blood test
- PPDM-C: patients with post-chronic pancreatitis diabetes mellitus
  Interventions: Diagnostic Test: blood test; Device: Continuous Glucose Monitor
- CP+IGT: patients with chronic pancreatitis combined with impaired glucose tolerance
  Interventions: Diagnostic Test: blood test; Device: Continuous Glucose Monitor
- CP+T2DM: patients with chronic pancreatitis combined with type 2 diabetes mellitus
  Interventions: Diagnostic Test: blood test; Device: Continuous Glucose Monitor

INTERVENTIONS:
Diagnostic Test: blood test — Evaluation of islets function and insulin secretion pattern： Evaluating the venous plasma glucose, c-peptide, and insulin concentrations at 0h, 0.5h, 1h, 2h, and 3h after the SBMT in patients with chronic pancreatitis.
  Characterization of pathophysiological features： Measuring intestinal hormones, exosomes, serum metabolites, and serum biochemical factors
Device: Continuous Glucose Monitor — blood glucose will be monitored 24 hours a day from 7 to 14 days by wearing continuous glucose monitor(only for patients who had new-onset diabetes or poor glycemic control )
  Groups: CP+IGT; CP+T2DM; PPDM-C

SUMMARY:
To evaluate the islet function and insulin secretion pattern of post-pancreatitis diabetes mellitus by oral glucose tolerance testing, and to explore the pathophysiological characteristics of PPDM-C which provide evidence for the diagnosis of PPDM-C.

DETAILED DESCRIPTION:
Blood samples will be collected from patients with chronic pancreatitis by oral glucose tolerance test (steamed bun meal test, SBMT) to assess their pancreatic islet function and insulin secretion pattern, measure other intestinal hormones, exosomes, plasma metabolites, and serum biochemical factors to characterize the pathophysiological features of PPDM-C and provide evidence for the diagnosis of PPDM-C. In order to better understand the glycemic fluctuations in patients with chronic pancreatitis combined with diabetes and guide subsequent treatment, Continuous Glucose Monitoring would be used in patients with chronic pancreatitis who had new-onset diabetes or poor glycemic control.

ELIGIBILITY:
Inclusion Criteria:

1. Age 15-85
2. patients with the diagnosis of chronic pancreatitis and diabetes mellitus (exclude type 1 diabetes).
3. participants with painless chronic pancreatitis were diagnosed with diabetes within 2 years of the diagnosis of chronic pancreatitis.
4. participants with painful chronic pancreatitis were diagnosed with diabetes after the first attack of chronic pancreatitis.
5. patients with chronic pancreatitis were previously diagnosed type 2 diabetes mellitus for more than 3 years.

Exclusion Criteria:

1. Participants with suspected malignant tumors of the pancreas or other sites of the body (including pancreatic cyst and Benign pancreatic tumor), or participants in the terminal stage of severe disease
2. Prior pancreatic surgery (including total pancreatectomy, pancreaticoduodenectomy, distal pancreatectomy, pancreatojejunostomy, or Frey), and prior bariatric or gastrointestinal surgery.
3. Serious mental illness, lesion of the liver (alanine aminotransferase or aspartate aminotransferase > 3 times the upper reference limit) or kidney (eGFR<60 mL/min/1.73 m2), pregnancy, breastfeeding or planning pregnancy, or accompanied with active liver diseases such as hepatitis B or hepatic cirrhosis.
4. Diagnosed type 1 diabetes, or other metabolic diseases that affect blood glucose
5. Using high-dose insulin preparations, or drugs affecting glucose metabolism (oral steroids, thiazide diuretics, beta-blockers, beta-agonist, nicotinic acid, immunosuppressant agents, antiretroviral drugs, and antipsychotics)
6. Acute complications of diabetes (diabetic ketoacidosis, severe hypoglycemia), severe microvascular disease (proliferative diabetic retinopathy, known diabetic nephropathy or neuropathy requiring treatment), and macrovascular disease (uncontrolled arterial hypertension, uncontrolled coronary artery disease, congestive heart failure, history of cerebrovascular event, seizure disorder, syncope, adrenal insufficiency, neurologic disease or atrial fibrillation) within the 12 months prior to enrollment.
7. Hospitalization for acute pancreatitis within the 2 months prior to enrollment or currently suffering acute inflammation.
8. Have been enrolled or currently participating in other clinical trials within the 3 months prior to enrollment.
9. Patients who refused to participate in the study

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic pancreatitis treated in the Department of Gastroenterology of Changhai Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
steamed bun meal test result 1 | Within 5 hours after the end of the steamed bread meal test
  Levels of glucose under the steamed bun meal experiment (100g flour made steamed bun)
steamed bun meal test result 2 | Within 6 hours after the end of the steamed bread meal test
  Levels of c-peptide bun meal experiment (100g flour made steamed bun)
steamed bun meal test result 3 | Within 7 hours after the end of the steamed bread meal test
  Levels of insulin under the steamed bun meal experiment (100g flour made steamed bun)

SECONDARY OUTCOMES:
gut hormone | up to 1 month
  Levels of gut hormone under the steamed bun meal experiment (100g flour made steamed bun)
Continuous glucose monitor results | after using continuous glucose monitor device for 7-14 days
  Time to target range (TIR) : the proportion of time with blood glucose fluctuation
glycemic control | at the time of enrollment
  glycosylated hemoglobin（%）

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, Changhai Hospital, Shanghai, Shanghai Municipality, China